CLINICAL TRIAL: NCT00151775
Title: Dose-ranging Study to Evaluate the Safety and Efficacy of Olmesartan Medoxomil in Children and Adolescents With Hypertension
Brief Title: Assessment of Efficacy and Safety of Olmesartan Medoxomil in Children and Adolescent Patients With High Blood Pressure
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS0866-A-U301
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Results first posted 2010-04-02 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-05

CONDITIONS: Hypertension
Keywords: Treatment of hypertension or high blood pressure in children ages 1-16 years.
MeSH Terms: conditions — Hypertension | interventions — Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Period 2 (Experimental): For Cohorts A and B, olmesartan medoxomil suspension 2.5 mg to 40 mg in patients 6-16 years old, depending on weight.
  For Cohort C, olmesartan medoxomil suspension 0.3 mg/kg to in patients 1-5 years old.
  Interventions: Drug: olmesartan medoxomil
- Period 3 (Experimental): Cohorts A, B, C - olmesartan medoxomil suspension or placebo taken once daily. Olmesartan medoxomil dose continued as in previous period.
  Interventions: Drug: olmesartan medoxomil; Drug: placebo
- Period 4 (Experimental): Cohorts A and B: Open label olmesartan medoxomil suspension or tablets 10mg - 40 mg
  Cohort C: Open label olmesartan medoxomil suspension 0.3 mg/kg - 0.6 mg/kg
  Interventions: Drug: olmesartan medoxomil

INTERVENTIONS:
Drug: olmesartan medoxomil — Cohorts A and B: 2.5mg to 40mg olmesartan, as a suspension (depending on weight), once daily. Tablets were used to prepare a suspension.
  Cohort C: 0.3mg/kg olmesartan ,as a suspension, once daily
  Other Names: Benicar (olmesartan medoxomil)
  Arms: Period 2; Period 3
Drug: placebo — Cohorts A, B, C: placebo, once daily
  Arms: Period 3
Drug: olmesartan medoxomil — Cohorts A and B: Open label olmesartan medoxomil suspension or tablets 10mg - 40 mg. Tablets were used to prepare the suspension or were given directly.
  Cohort C: Open label olmesartan medoxomil suspension 0.3 mg/kg - 0.6 mg/kg
  Other Names: Benicar (olmesartan medoxomil)
  Arms: Period 4

SUMMARY:
This study assesses the efficacy and safety of olmesartan medoxomil in children ages 1-16 with high blood pressure. After a 5-week blinded treatment period of up to 5 weeks participants can continue to take olmesartan medoxomil (OM) for up to an additional 46 weeks.

DETAILED DESCRIPTION:
This was a randomized, multicenter, double-blind, parallel-group, prospective dose-ranging study in subjects 1 to 16 years of age with hypertension. Subjects were enrolled into 1 of 3 cohorts based on age and race. Subjects 6 to 16 years of age were enrolled into Cohort A. Subjects enrolled into Cohort A were stratified by age with approximately half aged 6 to 12 years and the remainder aged 13 to 16 years. Approximately 15% of the subjects in Cohort A were to be Black or of African descent. When a minimum of 28 Black subjects were randomized into Cohort A, enrollment in Cohort B was started. Black subjects only, 6 to 16 years of age, were enrolled into Cohort B. For Cohorts A and B body weight of any patient was >=20Kg. Seated systolic blood pressure (SeSBP) was >=95th percentile for gender and height-for-age, or >=90th percentile if the patient is diabetic, or has glomerular kidney disease, or has a family history of hypertension. Patients with symptomatic hypertension requiring immediate established therapy, or who are above 2 standard deviations (SD) above the 99th percentile did not participate in the study.

Subjects 1 to 5 years of age were enrolled into Cohort C regardless of race. Body weight of any patient was >=5Kg. SeSBP was >=95th percentile for gender and height-for-age, or >=90th percentile if the patient is diabetic, or has glomerular kidney disease, or has a family history of hypertension. Patients on stable doses of concomitant antihypertensive agents including calcium channel blockers and/or diuretics only are permitted to enroll. Patients with symptomatic hypertension requiring immediate established therapy, or who are above 2 SD above the 99th percentile did not participate in the study.

The study comprised four periods. Period I was a wash-out period from Week -1 to randomization. Subjects were randomized to treatment sequences carried through the remainder of the study. Period II was a three-week, double-blind, dose-ranging period for Cohorts A and B, beginning at Day 1 and ending at the end of Week 3. In Cohorts A and B, subjects received either low-dose or high-dose olmesartan (OM) once daily. In Cohort C, Period II was an open-label OM treatment period where all subjects received 0.3 mg/kg OM per day. Period III was a double-blind, placebo-controlled withdrawal period beginning at Week 4 and ending after 1 or 2 weeks, depending on the seated blood pressure measurement at each weekly study visit. Subjects either continued their Period II OM regimen or switched to placebo based on the initial randomization scheme. Period IV was a 46-week open-label extension period.

ELIGIBILITY:
Inclusion Criteria:

* The patient's seated systolic BP (SeSBP) will be greater than or equal to 95th percentile for gender and height-for- age, or greater than or equal to 90th percentile if the patient is diabetic, or has glomerular kidney disease, or has a family history of hypertension.
* Negative for hepatitis B and C
* Negative for HIV

Exclusion Criteria:

* Patient should not have serious other conditions that could interfere with the analysis of the results or that could interfere with the well-being of the patient in the trial.
* Known sensitivity to olmesartan medoxomil
* Taking prohibited medication
* Consumed greater than 180 mg of caffeine daily
* Malignant hypertension
* History of congestive heart failure, cardiomyopathy, or obstructive valve disease
* Renal transplant within the previous 6 months
* Severe nephritic syndrome not in remission

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 362 (Actual)
Dates: Start 2005-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (65):
- United States (28):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Fresno, California
  - Los Angeles, California
  - Washington D.C., District of Columbia
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Decatur, Georgia
  - Honolulu, Hawaii
  - Park Ridge, Illinois
  - New Orleans, Louisiana
  - Shreveport, Louisiana
  - Baltimore, Maryland
  - Grand Rapids, Michigan
  - Las Vegas, Nevada
  - Hackensack, New Jersey
  - New Brunswick, New Jersey
  - Kinston, North Carolina
  - Cincinnati, Ohio
  - Dayton, Ohio
  - Portland, Oregon
  - Beaumont, Texas
  - Houston, Texas
  - Charlottesville, Virginia
- Argentina (5):
  - San Miguel de Tucumán, TUC
  - Bahía Blanca
  - Buenos Aires
  - Capital Federal
  - Mar del Plata
- Brazil (5):
  - Campinas
  - Curitiba
  - Porto Alegre
  - Recife
  - São Paulo
- Santiago, Chile
- Colombia (2):
  - Bogotá
  - Cali-Valle
- India (9):
  - Ahmedabad, Gujarat
  - Mangalore, Karna
  - Vellore, Karna
  - Trivandrum, Kerala
  - Lucknow, Uttar Prad
  - Chandigarh
  - Hyderabad
  - New Delhi
  - Tamil Nadu
- Nairobi, Kenya
- Lima, Peru
- South Africa (10):
  - Bloemfontein
  - Cape Town
  - Durban, KZ-Natal
  - E Cape
  - Eastern Cape
  - Park Town, Gauteng
  - Pietermaritzburg, KZ-Natal
  - Potchefstroom, Northwest
  - Pretoria, Gauteng
  - Western Cape
- Kampala, Uganda
- Zambia (2):
  - Kitwe
  - Lusaka

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Period 1 was a screening, wash-out period of approximately two weeks. All participants were included in the screening, wash-out period and during this period no intervention was administered.
Groups:
- Cohort A: High Dose OM in Periods 2, 3: Subgroup of Cohort A (6-16 years old with a limit on the number of Black participants) given a high dose (20 mg or 40 mg) of olmesartan medoxomil suspension (OM) depending on weight during Period 2 (double-blind, dose-response period from day 0 to week 3). Half of the participants continued this dose into Period 3 (double-blind, placebo controlled period from week 3 to week 5).
- Cohort A: Low Dose OM in Periods 2, 3: Subgroup of Cohort A (6-16 years old with a limit on the number of Black participants) given a low dose (2.5 mg or 5.0 mg) of olmesartan medoxomil suspension (OM) depending on weight during Period 2 (double-blind, dose-response period from day 0 to week 3). Half of the participants continued this dose into Period 3 (double-blind, placebo controlled period from week 3 to week 5).
- Cohort A: Placebo in Period 3 (From High Dose in Period 2): Subgroup of Cohort A (6-16 years old with a limit on the number of Black participants) given placebo during Period 3 (double-blind, placebo-controlled period from week 3 to week 5) instead of the previous high dose of olmesartan
- Cohort A: Placebo in Period 3 (From Low Dose in Period 2): Subgroup of Cohort A (6-16 years old with a limit on the number of Black participants) given placebo during Period 3 (double-blind, placebo-controlled period from week 3 to week 5) instead of the previous low dose of olmesartan.
- Cohort A: Period 4 Open-label OM: All members of Cohort A (6-16 years old with a limit on the number of Black participants) were given 10 mg to 40 mg of olmesartan (OM) administered as oral suspension or tablets depending on participant weight and response in the open-label Period 4 (weeks 6-51). Additional antihypertensive drugs (not an angiotensin converting enzyme or angiotensin receptor blocker) were allowed if hypertension was not controlled.
- Cohort B: High Dose OM in Periods 2, 3: Subgroup of Cohort B (6-16 years old comprised exclusively of Black participants) given a high dose (20 mg or 40 mg) of olmesartan medoxomil suspension (OM) depending on weight during Period 2 (double-blind, dose-response period from day 0 to week 3). Half of the participants continued this dose into Period 3 (double-blind, placebo controlled period from week 3 to week 5).
- Cohort B: Low Dose OM in Periods 2, 3: Subgroup of Cohort B (6-16 years old comprised exclusively of Black participants) given a low dose (2.5 mg or 5.0 mg) of olmesartan medoxomil suspension (OM) depending on weight during Period 2 (double-blind, dose-response period from day 0 to week 3). Half of the participants continued this dose into Period 3 (double-blind, placebo controlled period from week 3 to week 5).
- Cohort B: Placebo in Period 3 (From High Dose in Period 2): Subgroup of Cohort B (6-16 years old comprised exclusively of Black participants) given placebo during Period 3 (double-blind, placebo-controlled period from week 3 to week 5) instead of the previous high dose of olmesartan.
- Cohort B: Placebo in Period 3 (From Low Dose in Period 2): Subgroup of Cohort B (6-16 years old comprised exclusively of Black participants) given placebo during Period 3 (double-blind, placebo-controlled period from week 3 to week 5) instead of the previous low dose of olmesartan.
- Cohort B: Period 4 Open-label OM: All members of Cohort B (6-16 years old comprised exclusively of Black participants) were given 10 mg to 40 mg of olmesartan (OM) administered as oral suspension or tablets depending on participant weight and response in the open-label Period 4 (weeks 6-51). Additional antihypertensive drugs (not an angiotensin converting enzyme or angiotensin receptor blocker) were allowed if hypertension was not controlled.
- Cohort C: OM in Periods 2, 3, 4: Cohort C (1-5 years old) was given olmesartan medoxomil (OM) 0.3 mg/kg in Period 2 (open-label period from day 0 to week 3) and a subgroup of Cohort C was given that dose of OM during Period 3 (double-blind, placebo-controlled period from week 3 to week 5). In Period 4 (open-label period from weeks 6-51), all of Cohort C received an OM starting dose of 0.3 mg/kg. If hypertension was not controlled after two week the dose was doubled. Additional antihypertensive drugs (not an angiotensin converting enzyme or angiotensin receptor blocker) were allowed if hypertension was not controlled.
- Cohort C: Placebo in Period 3 (From OM in Period 2): Subgroup of Cohort C (1-5 years old) given placebo during Period 3 (double-blind, placebo-controlled period from week 3 to week 5).
Period: Period 2 - Double-Blind Dose Response
Arm/Group | Cohort A: High Dose OM in Periods 2, 3 | Cohort A: Low Dose OM in Periods 2, 3 | Cohort A: Placebo in Period 3 (From High Dose in Period 2) | Cohort A: Placebo in Period 3 (From Low Dose in Period 2) | Cohort A: Period 4 Open-label OM | Cohort B: High Dose OM in Periods 2, 3 | Cohort B: Low Dose OM in Periods 2, 3 | Cohort B: Placebo in Period 3 (From High Dose in Period 2) | Cohort B: Placebo in Period 3 (From Low Dose in Period 2) | Cohort B: Period 4 Open-label OM | Cohort C: OM in Periods 2, 3, 4 | Cohort C: Placebo in Period 3 (From OM in Period 2)
Started | 95 | 95 | 0 | 0 | 0 | 56 | 56 | 0 | 0 | 0 | 60 | 0
Completed | 93 | 89 | 0 | 0 | 0 | 54 | 53 | 0 | 0 | 0 | 59 | 0
Not Completed | 2 | 6 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — non-compliance | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — The blood pressure goal was met | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Period 3: Double-blind, Withdrawal
Arm/Group | Cohort A: High Dose OM in Periods 2, 3 | Cohort A: Low Dose OM in Periods 2, 3 | Cohort A: Placebo in Period 3 (From High Dose in Period 2) | Cohort A: Placebo in Period 3 (From Low Dose in Period 2) | Cohort A: Period 4 Open-label OM | Cohort B: High Dose OM in Periods 2, 3 | Cohort B: Low Dose OM in Periods 2, 3 | Cohort B: Placebo in Period 3 (From High Dose in Period 2) | Cohort B: Placebo in Period 3 (From Low Dose in Period 2) | Cohort B: Period 4 Open-label OM | Cohort C: OM in Periods 2, 3, 4 | Cohort C: Placebo in Period 3 (From OM in Period 2)
Started | 48 | 45 | 45 | 44 | 0 | 26 | 27 | 28 | 26 | 0 | 29 | 29
Completed | 48 | 45 | 42 | 44 | 0 | 25 | 26 | 27 | 26 | 0 | 29 | 28
Not Completed | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Met blood pressure goal | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 4: Open Label
Arm/Group | Cohort A: High Dose OM in Periods 2, 3 | Cohort A: Low Dose OM in Periods 2, 3 | Cohort A: Placebo in Period 3 (From High Dose in Period 2) | Cohort A: Placebo in Period 3 (From Low Dose in Period 2) | Cohort A: Period 4 Open-label OM | Cohort B: High Dose OM in Periods 2, 3 | Cohort B: Low Dose OM in Periods 2, 3 | Cohort B: Placebo in Period 3 (From High Dose in Period 2) | Cohort B: Placebo in Period 3 (From Low Dose in Period 2) | Cohort B: Period 4 Open-label OM | Cohort C: OM in Periods 2, 3, 4 | Cohort C: Placebo in Period 3 (From OM in Period 2)
Started | 0 | 0 | 0 | 0 | 179 | 0 | 0 | 0 | 0 | 104 | 57 | 0
Completed | 0 | 0 | 0 | 0 | 149 | 0 | 0 | 0 | 0 | 83 | 57 | 0
Not Completed | 0 | 0 | 0 | 0 | 30 | 0 | 0 | 0 | 0 | 21 | 0 | 0
Not completed — Increased blood pressure | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 7 | 0 | 0
Not completed — Non-compliance with protocol | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 4 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort A: High Dose OM: Subgroup of Cohort A (6-16 years old with a limit on the number of Black participants) given a high dose (20 mg or 40 mg) of olmesartan medoxomil suspension (OM) depending on weight during Period 2 (double-blind, dose-response period). Half of the participants continued this dose into Period 3 (double-blind, placebo controlled period).
- Cohort A: Low Dose OM: Subgroup of Cohort A (6-16 years old with a limit on the number of Black participants) given a low dose (2.5 mg or 5.0 mg) of olmesartan medoxomil suspension (OM) depending on weight during Period 2 (double-blind, dose-response period). Half of the participants continued this dose into Period 3 (double-blind, placebo controlled period).
- Cohort B: High Dose OM: Subgroup of Cohort B (6-16 years old comprised exclusively of Black participants) given a high dose (20 mg or 40 mg) of olmesartan medoxomil suspension (OM) depending on weight during Period 2 (double-blind, dose-response period). Half of the participants continued this dose into Period 3 (double-blind, placebo controlled period).
- Cohort B: Low Dose OM: Subgroup of Cohort B (6-16 years old comprised exclusively of Black participants) given a low dose (2.5 mg or 5.0 mg) of olmesartan medoxomil suspension (OM) depending on weight during Period 2 (double-blind, dose-response period). Half of the participants continued this dose into Period 3 (double-blind, placebo controlled period).
- Cohort C: OM (Olmesartan Medoxomil): Cohort C (1-5 years old) was given olmesartan medoxomil (OM) 0.3 mg/kg in Period 2 (open-label period) and a subgroup of Cohort C was given that dose of OM during Period 3 (double-blind, placebo-controlled period). In Period 4 (open-label period), all of Cohort C received an OM starting dose of 0.3 mg/kg. If hypertension was not controlled after two week the dose was doubled. Additional antihypertensive drugs (not an angiotensin converting enzyme or angiotensin receptor blocker) were allowed if hypertension was not controlled.
- Total: Total of all reporting groups
Arm/Group | Cohort A: High Dose OM | Cohort A: Low Dose OM | Cohort B: High Dose OM | Cohort B: Low Dose OM | Cohort C: OM (Olmesartan Medoxomil) | Total
Number analyzed (Participants) | 95 | 95 | 56 | 56 | 60 | 362
Age, Continuous [Mean (Standard Deviation); unit: years] — The data provided for the total study population includes only Cohorts A+B.
  years | 12.1 (2.97) | 12.3 (2.98) | 12.2 (2.83) | 12.8 (2.42) | 3.4 (1.45) | 12.3 (2.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 35 | 35 | 20 | 26 | 149
  Male | 62 | 60 | 21 | 36 | 34 | 213
Race/Ethnicity, Customized [Number; unit: Participants]
  Latino/Hispanic | 42 | 47 | 0 | 1 | 27 | 117
  non-Latino/Hispanic | 53 | 48 | 56 | 55 | 33 | 245
Height [Mean (Standard Deviation); unit: cm] — The data provided for the total study population is only for Cohorts A+B
  cm | 153.3 (18.46) | 155.1 (19.12) | 154.2 (17.83) | 156.1 (14.21) | 98.3 (12.92) | 154.6 (17.79)
Seated Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] — The data provided for the total study population is only for Cohort A+B
  mm Hg | 129.1 (8.32) | 129.5 (9.10) | 130.8 (9.73) | 131.7 (9.12) | 115.2 (8.74) | 130.0 (9.00)
Seated diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] — The data provided for the total study population consists only of Cohort A+B
  mm Hg | 76.3 (8.09) | 78.1 (8.17) | 79.2 (7.08) | 79.4 (9.05) | 72.7 (8.74) | 78.0 (8.18)
Weight [Mean (Standard Deviation); unit: kg] — The data provided for the total study population is only for Cohort A+B
  kg | 68.0 (34.22) | 78.9 (41.85) | 66.2 (32.39) | 68.1 (34.36) | 16.9 (6.61) | 71.1 (36.72)

OUTCOME MEASURES:

1. Primary Outcome: Least Squares Mean Change From Baseline in Seated Systolic Blood Pressure to the End of Period 2 (3 Weeks)
Description: The efficacy dose response change in trough seated systolic blood pressure (both non-weight adjusted and weight adjusted results) from baseline to the end of the dose-ranging period (Period 2). Non-weight adjusted dose was the fixed olmesartan medoxomil dose; weight adjusted dose calculated mg of olmesartan medoxomil per kg of weight at baseline.
Time Frame: Day 0 to 3 weeks
Population: The number of participants includes all randomized to Cohort A, Cohort B and a combination of the two cohorts. The Last Observation Carried Forward method was used in the linear regression analysis for the change in the seated systolic blood pressure from baseline to the end of three weeks.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Groups:
- Cohort A: Cohort A participants were 6-16 years old with a limit on the number of Black participants. Includes participants randomized to both the high dose of olmesartan medoxomil suspension (20 mg or 40 mg) and the low dose (2.5 mg or 5.0mg), depending on weight, administered once daily.
- Cohort B: Cohort B participants were 6-16 years old and comprised exclusively of Black participants. Includes participants randomized to both the high dose of olmesartan medoxomil suspension (20 mg or 40 mg) and the low dose (2.5 mg or 5.0 mg), depending on weight, administered once daily.
- Cohorts A + B: Cohort A + B participants were 6-16 years old. Cohort A limited the number of Black participants, while Cohort B was comprised exclusively of Black participants. Includes participants randomized to both the high dose of olmesartan medoxomil suspension (20 mg or 40 mg) and the low dose (2.5 mg or 5.0mg), depending on weight, administered once daily.
Arm/Group | Cohort A | Cohort B | Cohorts A + B
Number analyzed (Participants) | 190 | 112 | 302
mm Hg
  Non-weight adjusted dosage | -0.69 (0.202) | -0.85 (0.282) | -0.75 (0.165)
  Weight adjusted dosage | -8.97 (2.054) | -7.17 (3.190) | -8.36 (1.750)
Statistical Analysis 1: Comparison: Cohort A; Non-weight adjusted dosage; Test type: Superiority or Other; p = 0.0008, Regression, Linear
Statistical Analysis 2: Comparison: Cohort A; Weight adjusted dosage; Test type: Superiority or Other; p < 0.0001, Regression, Linear
Statistical Analysis 3: Comparison: Cohort B; Non-weight adjusted dosage; Test type: Superiority or Other; p = 0.0032, Regression, Linear
Statistical Analysis 4: Comparison: Cohort B; Weight adjusted dosage; Test type: Superiority or Other; p = 0.0265, Regression, Linear
Statistical Analysis 5: Comparison: Cohorts A + B; Non-weight adjusted dosage; Test type: Superiority or Other; p < 0.0001, Regression, Linear
Statistical Analysis 6: Comparison: Cohorts A + B; Weight adjusted dosage; Test type: Superiority or Other; p < 0.0001, Regression, Linear

2. Primary Outcome: Mean Change From Baseline in Seated Systolic and Diastolic Blood Pressure Measurements to the End of Period 2 (3 Weeks)
Description: Mean change from baseline to the end of the dose ranging period in systolic and diastolic blood pressure readings for Cohort A, Cohort B and Cohorts A+B combined.
Time Frame: Day 0 (baseline) to 3 weeks
Population: The Intent-to-Treat (ITT) population for Period II of the study was defined as subjects who took at least one dose of study medication and had study baseline and at least one seated systolic, or diastolic blood pressure measurement after taking study medication. The Last Observation carried forward was used
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Cohorts A + B: Low Dose OM: Subgroup from Cohorts A + B (6-16 years old) who received the low dose of olmesartan medoxomil suspension (OM 2.5 mg or 5.0 mg depending on weight), administered once daily in Period 2. Cohort A limited the number of Black participants, while Cohort B was comprised exclusively of Black participants.
- Cohorts A + B: High Dose OM: Subgroup from Cohorts A + B (6-16 years old) who received the high dose of olmesartan medoxomil suspension (OM 20 mg or 40 mg depending on weight), administered once daily in Period 2. Cohort A limited the number of Black participants, while Cohort B was comprised exclusively of Black participants.
Arm/Group | Cohort A: Low Dose OM | Cohort A: High Dose OM | Cohort B: Low Dose OM | Cohort B: High Dose OM | Cohorts A + B: Low Dose OM | Cohorts A + B: High Dose OM
Number analyzed (Participants) | 94 | 94 | 56 | 56 | 150 | 150
mm Hg
  Change in Systolic Blood Pressure | -7.76 (9.180) | -12.58 (10.157) | -4.73 (11.483) | -10.68 (9.259) | -6.63 (10.170) | -11.87 (9.843)
  Change in Diastolic Blood Pressure | -5.52 (8.058) | -9.50 (9.757) | -3.49 (8.844) | -7.58 (8.172) | -4.76 (8.389) | -8.78 (9.216)
Statistical Analysis 1: Comparison: Cohort A: Low Dose OM vs Cohort A: High Dose OM; A linear regression analysis of olmesartan dose (non-weight adjusted) on the change from baseline in seated systolic blood pressure was carried out. The null hypothesis of zero-slope was tested; Test type: Superiority or Other; p = 0.0008, Regression, Linear; Slope = 0.69
Statistical Analysis 2: Comparison: Cohort A: Low Dose OM vs Cohort A: High Dose OM; A linear regression analysis of olmesartan dose (non-weight adjusted) on the change from baseline in seated diastolic blood pressure was carried out. The null hypothesis of zero-slope was tested; Test type: Superiority or Other; p = 0.0026, Regression, Linear; Slope = -.057
Statistical Analysis 3: Comparison: Cohort B: Low Dose OM vs Cohort B: High Dose OM; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0032, Regression, Linear; Slope = -0.85
Statistical Analysis 4: Comparison: Cohort B: Low Dose OM vs Cohort B: High Dose OM; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p = 0.0125, Regression, Linear; Slope = -0.58
Statistical Analysis 5: Comparison: Cohorts A + B: Low Dose OM vs Cohorts A + B: High Dose OM; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Linear; Slope = -0.75
Statistical Analysis 6: Comparison: Cohorts A + B: Low Dose OM vs Cohorts A + B: High Dose OM; [analysis description as in outcome 2, analysis 2]; Test type: Superiority or Other; p < 0.0001, Regression, Linear; Slope = -0.57
Statistical Analysis 7: Comparison: Cohort A: Low Dose OM vs Cohort A: High Dose OM; A linear regression analysis of olmesartan dose (weight adjusted) on the change from baseline in seated systolic blood pressure was carried out. The null hypothesis of zero-slope was tested; Test type: Superiority or Other; p < 0.0001, Regression, Linear; Slope = -8.97
Statistical Analysis 8: Comparison: Cohort A: Low Dose OM vs Cohort A: High Dose OM; A linear regression analysis of olmesartan dose (weight adjusted) on the change from baseline in seated diastolic blood pressure was carried out. The null hypothesis of zero-slope was tested; Test type: Superiority or Other; p < 0.0001, Regression, Linear; Slope = -8.15
Statistical Analysis 9: Comparison: Cohort B: Low Dose OM vs Cohort B: High Dose OM; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p = 0.0265, Regression, Linear; Slope = -7.17
Statistical Analysis 10: Comparison: Cohort B: Low Dose OM vs Cohort B: High Dose OM; [analysis description as in outcome 2, analysis 8]; Test type: Superiority or Other; p = 0.0084, Regression, Linear; Slope = -6.85
Statistical Analysis 11: Comparison: Cohorts A + B: Low Dose OM vs Cohorts A + B: High Dose OM; [analysis description as in outcome 2, analysis 7]; Test type: Superiority or Other; p < 0.0001, Regression, Linear; Slope = -8.36
Statistical Analysis 12: Comparison: Cohorts A + B: Low Dose OM vs Cohorts A + B: High Dose OM; [analysis description as in outcome 2, analysis 8]; Test type: Superiority or Other; p < 0.0001, Regression, Linear; Slope = -7.71

3. Secondary Outcome: Mean Change From Period 3 Baseline in Seated Systolic and Diastolic Blood Pressure Measurements to the End of Period 3
Description: Mean change from period 3 baseline (completion of the dose adjustment period and prior to starting the treatment of period 3) to the end of period 3 (double-blind placebo-controlled period) in seated systolic and diastolic blood pressure readings for Cohort A, Cohort B and Cohorts A+B combined.
Time Frame: Week 3 (period 3 baseline) to week 5 (end of Period 3)
Population: Intent to treat population defined as subjects who finished Period 2, had the end of Period 2 seated systolic or diastolic blood pressure measurement, took the Period 3 study medication for at least one week, and had the end of Period 3 seated systolic or diastolic blood pressure measurement.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Cohort A: OM Period 3: Cohort A participants were 6-16 years old with a limit on the number of Black participants. Includes participants randomized to both the high dose of olmesartan medoxomil suspension (OM 20 mg or 40 mg) and the low dose (2.5 mg or 5.0mg), depending on weight, administered once daily in period 2, and continued that dosage into period 3.
- Cohort A: Placebo Period 3: Cohort A participants were 6-16 years old with a limit on the number of Black participants. Includes participants randomized to both the high and low dose of olmesartan medoxomil suspension in period 2, and changed to placebo in period 3.
- Cohort B: OM Period 3: Cohort B participants were 6-16 years old and comprised exclusively of Black participants. Includes participants randomized to both the high dose of olmesartan medoxomil suspension (OM 20 mg or 40 mg) and the low dose (2.5 mg or 5.0mg), depending on weight, administered once daily in period 2, and continued that dosage into period 3.
- Cohort B: Placebo Period 3: Cohort B participants were 6-16 years old and comprised exclusively of Black participants. Includes participants randomized to both the high and low dose of olmesartan medoxomil suspension in period 2, and changed to placebo in period 3.
- Cohorts A + B: OM Period 3: Cohort A + B participants were 6-16 years old. Includes participants randomized to both the high dose of olmesartan medoxomil suspension (OM 20 mg or 40 mg) and the low dose (2.5 mg or 5.0mg), depending on weight, administered once daily in period 2, and continued that dosage into period 3.
- Cohorts A + B: Placebo Period 3: Cohorts A + B participants were 6-16 years old. Includes participants randomized to both the high and low dose of olmesartan medoxomil suspension in period 2, and changed to placebo in period 3.
Arm/Group | Cohort A: OM Period 3 | Cohort A: Placebo Period 3 | Cohort B: OM Period 3 | Cohort B: Placebo Period 3 | Cohorts A + B: OM Period 3 | Cohorts A + B: Placebo Period 3
Number analyzed (Participants) | 93 | 89 | 53 | 54 | 146 | 143
mm Hg
  Change in Systolic Blood Pressure | 0.43 (9.46) | 4.93 (9.62) | 1.37 (9.50) | 3.79 (10.00) | 0.77 (9.451) | 4.50 (9.745)
  Change in Diastolic Blood Pressure | 0.24 (8.12) | 4.43 (10.15) | 1.94 (7.10) | 3.25 (8.74) | 0.85 (7.790) | 3.99 (9.627)
Statistical Analysis 1: Comparison: Cohort A: OM Period 3 vs Cohort A: Placebo Period 3; Analysis of systolic blood pressure. Null hypothesis of no treatment difference was tested; Test type: Superiority or Other; p = 0.0093, ANCOVA; The ANCOVA model used treatment and country as fixed effects and baseline as covariate; LS Mean Difference = -3.58, 95% CI 2-sided [-6.27 to -0.89]
Statistical Analysis 2: Comparison: Cohort A: OM Period 3 vs Cohort A: Placebo Period 3; Analysis for diastolic blood pressure. The null hypothesis of no treatment difference was tested; Test type: Superiority or Other; p = 0.0052, ANCOVA; The ANCOVA model used treatment and country as fixed effects and baseline as covariate; LS Mean difference = -3.49, 95% CI 2-sided [-5.92 to -1.05]
Statistical Analysis 3: Comparison: Cohort B: OM Period 3 vs Cohort B: Placebo Period 3; Analysis of systolic blood pressure. Null hypothesis of no treatment difference was tested; Test type: Superiority or Other; p = 0.1330, ANCOVA; The ANCOVA model used treatment and country as fixed effects and baseline as covariate; LS Mean difference = -2.57, 95% CI 2-sided [-5.93 to 0.79]
Statistical Analysis 4: Comparison: Cohort B: OM Period 3 vs Cohort B: Placebo Period 3; Analysis for diastolic blood pressure. The null hypothesis of no treatment difference was tested; Test type: Superiority or Other; p = 0.3442, ANCOVA; The ANCOVA model used treatment and country as fixed effects and baseline as covariate; LS Mean difference = -1.38, 95% CI 2-sided [-4.27 to 1.50]
Statistical Analysis 5: Comparison: Cohorts A + B: OM Period 3 vs Cohorts A + B: Placebo Period 3; For seated systolic blood pressure the null hypothesis of no treatment difference was tested; Test type: Superiority or Other; p = 0.0029, ANCOVA; The ANCOVA model used treatment and country as fixed effects and baseline as covariate; LS Mean difference = -3.16, 95% CI 2-sided [-5.24 to -1.09]
Statistical Analysis 6: Comparison: Cohorts A + B: OM Period 3 vs Cohorts A + B: Placebo Period 3; For seated diastolic blood pressure the null hypothesis of no treatment difference was tested; Test type: Superiority or Other; p = 0.0032, ANCOVA; The ANCOVA model used treatment and country as fixed effects and baseline as covariate; LS Mean difference = -2.80, 95% CI 2-sided [-4.65 to -0.95]

4. Secondary Outcome: Mean Change From Period 3 Baseline in Seated Systolic and Diastolic Blood Pressure Measurements to the End of Period 3
Description: Mean change from period 3 baseline (completion of the dose adjustment period and prior to starting the treatment of period 3) to the end of period 3 (double-blind placebo-controlled period) in seated systolic and diastolic blood pressure readings for Cohort C.
Time Frame: Week 3 (period 3 baseline) to week 5 (end of Period 3)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Cohort C: OM Period 3: Cohort C consisted of children from 1 to 5 years of age. There were no racial restrictions. This group continued on its Period 2 olmesartan dose of 0.3 mg/kg.
- Cohort C: Placebo Period 3: Cohort C consisted of children from 1 to 5 years of age. There were no racial restrictions. This group was switched from its Period 2 olmesartan dose of 0.3 mg/kg to placebo.
Arm/Group | Cohort C: OM Period 3 | Cohort C: Placebo Period 3
Number analyzed (Participants) | 29 | 29
mm Hg
  Seated Systolic Blood Pressure | 1.36 (8.994) | 4.95 (8.568)
  Seated Diastolic Blood Pressure | 0.31 (8.556) | 3.77 (7.203)
Statistical Analysis 1: Comparison: Cohort C: OM Period 3 vs Cohort C: Placebo Period 3; For seated systolic blood pressure the null hypothesis of no treatment difference was tested; Test type: Superiority or Other; p = 0.2113, ANCOVA; The ANCOVA model used treatment and country as fixed effects and baseline as covariate; LS Mean difference = -2.82, 95% CI 2-sided [-7.29 to 1.65]
Statistical Analysis 2: Comparison: Cohort C: OM Period 3 vs Cohort C: Placebo Period 3; For seated diastolic blood pressure the null hypothesis of no treatment difference was tested; Test type: Superiority or Other; p = 0.1496, ANCOVA; The ANCOVA model used treatment and country as fixed effects and baseline as covariate; LS Mean difference = -2.92, 95% CI 2-sided [-6.92 to 1.09]

5. Secondary Outcome: Mean Change From Baseline in Seated Systolic and Diastolic Blood Pressure Measurements to the End of Period 4 (End of Study)
Description: Mean change from baseline to the end of the open label Period 4 in seated systolic and diastolic blood pressure readings for Cohort A, Cohort B and Cohorts A+B combined.
Time Frame: Day 0 to week 51 (end of study)
Population: Intent to treat population includes participants with at least one visit in Period 4.
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Cohort A: Period 4 Open-label OM: All members of Cohort A (6-16 years old with a limit on the number of Black participants) were given 10 mg to 40 mg of olmesartan (OM) administered as oral suspension or tablets depending on participant weight and response in the open-label Period 4. Additional antihypertensive drugs (not an angiotensin converting enzyme or angiotensin receptor blocker) were allowed if hypertension was not controlled.
- Cohort B: Period 4 Open-label OM: All members of Cohort B (6-16 years old comprised exclusively of Black participants) were given 10 mg to 40 mg of olmesartan (OM) administered as oral suspension or tablets depending on participant weight and response in the open-label Period 4. Additional antihypertensive drugs (not an angiotensin converting enzyme or angiotensin receptor blocker) were allowed if hypertension was not controlled.
- Cohorts A + B: Period 4 Open-label OM: All members of Cohorts A + B (6-16 years old) were given 10 mg to 40 mg of olmesartan (OM) administered as oral suspension or tablets depending on participant weight and response in the open-label Period 4. Additional antihypertensive drugs (not an angiotensin converting enzyme or angiotensin receptor blocker) were allowed if hypertension was not controlled.
Arm/Group | Cohort A: Period 4 Open-label OM | Cohort B: Period 4 Open-label OM | Cohorts A + B: Period 4 Open-label OM
Number analyzed (Participants) | 178 | 103 | 281
mm Hg
  Change in Systolic Blood Pressure | -10.8 (9.75) | -7.7 (12.71) | -9.7 (11.01)
  Change in Diastolic Blood Pressure | -7.4 (9.31) | -5.1 (9.45) | -6.6 (9.41)

6. Secondary Outcome: Mean Change From Baseline in Seated Systolic and Diastolic Blood Pressure Measurements to the End of Period 4 (End of Study)
Description: Mean change from baseline to the end of the open label Period 4 in seated systolic and diastolic blood pressure readings for Cohort C.
Time Frame: Day 0 to week 51 week (end of study)
Population: 57=the number of participants who received medication in Period 4
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Cohort C: OM (Olmesartan Medoxomil)
Number analyzed (Participants) | 57
mm Hg
  Change in Systolic Blood Pressure | -15.7 (9.83)
  Change in Diastolic Blood Pressure | -13.3 (11.18)

ADVERSE EVENTS:
Time Frame: Adverse events were collected starting with the signing of the informed consent form and continuing through the end of the study (51 weeks)
Description: AEs observed by the investigator, or reported by the subject, and any remedial action taken, were recorded in the case report form by the investigator. The nature of each event, time of onset after drug administration, duration, and intensity were documented together with the investigator's opinion of the causal relationship to the treatment.
Groups:
- Cohort A: Period 2 High Dose OM; Cohort B: Period 2 High Dose OM: For Cohort A (participants 6-16 years old), olmesartan medoxomil suspension (OM) providing 20 mg or 40 mg, depending on weight.
- Cohort A: Period 2 Low Dose OM: For Cohort A (participants 6-16 years old), olmesartan medoxomil suspension (OM) providing 2.5 mg or 5 mg, depending on weight.
- Cohort A: Period 3 OM High Dose Continued; Cohort B: Period 3 OM High Dose Continued: The 20 mg or 40 mg dose of olmesartan medoxomil suspension (OM) from the previous period was continued.
- Cohort A: Period 3 Placebo From High Dose; Cohort B: Period 3 Placebo From High Dose: Placebo was given instead of the previous high dose of olmesartan
- Cohort A: Period 3 OM Low Dose Continued; Cohort B: Period 3 OM Low Dose Continued: The 2.5 mg or 5 mg dose of olmesartan medoxomil suspension (OM) from the previous period was continued.
- Cohort A: Period 3 Placebo From Low Dose; Cohort B: Period 3 Placebo From Low Dose: Placebo was given instead of the previous low dose of olmesartan
- Cohort A: Period 4 Open-label OM: 10 mg to 40 mg of olmesartan (OM) was administered as oral suspension or tablets depending on participant weight and response. Additional antihypertensive drugs (not an angiotensin converting enzyme or angiotensin receptor blocker) were allowed if hypertension was not controlled.
- Cohort B: Period 2 Low Dose OM: For Cohort B (participants 6-16 years old), olmesartan medoxomil suspension (OM) providing 2.5 mg or 5 mg, depending on weight.
- Cohort B: Period 4 Open-label OM: 10 mg to 40 mg of olmesartan (OM) was administered as oral suspension or tablets depending on particpant weight and response. Additional antihypertensive drugs (not an angiotensin converting enzyme or angiotensin receptor blocker) were allowed if hypertension was not controlled.
- Cohort C: Period 2 Open-label OM: The dose of olmesartan medoxomil suspension (OM) was 0.3 mg/kg for all particpants who were 1 to 5 years of age.
- Cohort C: Period 3 OM Dose Continued: The 0.3 mg/kg dose of OM was continued for these participants
- Cohort C: Period 3 Placebo: The 0.3 mg/kg dose of olmesartan medoxomil suspension (OM) was discontinued for these participants. They were switched to placebo.
- Cohort C: Period 4 Open-label OM: Participants received an olmesartan medoxomil suspension (OM) starting dose of 0.3 mg/kg. If hypertension was not controlled after two week the dose was doubled. Additional antihypertensive drugs (not an angiotensin converting enzyme or angiotensin receptor blocker) were allowed if hypertension was not controlled.
Arm/Group | Cohort A: Period 2 High Dose OM | Cohort A: Period 2 Low Dose OM | Cohort A: Period 3 OM High Dose Continued | Cohort A: Period 3 Placebo From High Dose | Cohort A: Period 3 OM Low Dose Continued | Cohort A: Period 3 Placebo From Low Dose | Cohort A: Period 4 Open-label OM | Cohort B: Period 2 High Dose OM | Cohort B: Period 2 Low Dose OM | Cohort B: Period 3 OM High Dose Continued | Cohort B: Period 3 Placebo From High Dose | Cohort B: Period 3 OM Low Dose Continued | Cohort B: Period 3 Placebo From Low Dose | Cohort B: Period 4 Open-label OM | Cohort C: Period 2 Open-label OM | Cohort C: Period 3 OM Dose Continued | Cohort C: Period 3 Placebo | Cohort C: Period 4 Open-label OM
Serious Adverse Events (participants affected / at risk) | 2/95 | 1/95 | 0/48 | 0/45 | 0/45 | 0/44 | 20/179 | 0/56 | 0/56 | 1/26 | 0/28 | 0/27 | 0/26 | 7/104 | 0/59 | 0/29 | 0/29 | 6/57
Other Adverse Events (participants affected / at risk) | 47/95 | 46/95 | 15/48 | 6/45 | 9/45 | 6/44 | 128/178 | 9/56 | 12/56 | 4/26 | 1/28 | 2/27 | 1/26 | 56/103 | 12/59 | 4/29 | 8/28 | 46/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Cohort A: Period 2 High Dose OM (N=95) | Cohort A: Period 2 Low Dose OM (N=95) | Cohort A: Period 3 OM High Dose Continued (N=48) | Cohort A: Period 3 Placebo From High Dose (N=45) | Cohort A: Period 3 OM Low Dose Continued (N=45) | Cohort A: Period 3 Placebo From Low Dose (N=44) | Cohort A: Period 4 Open-label OM (N=179) | Cohort B: Period 2 High Dose OM (N=56) | Cohort B: Period 2 Low Dose OM (N=56) | Cohort B: Period 3 OM High Dose Continued (N=26) | Cohort B: Period 3 Placebo From High Dose (N=28) | Cohort B: Period 3 OM Low Dose Continued (N=27) | Cohort B: Period 3 Placebo From Low Dose (N=26) | Cohort B: Period 4 Open-label OM (N=104) | Cohort C: Period 2 Open-label OM (N=59) | Cohort C: Period 3 OM Dose Continued (N=29) | Cohort C: Period 3 Placebo (N=29) | Cohort C: Period 4 Open-label OM (N=57)
Abcess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anasarca (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Broncopneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2
Coarctation of the aorta (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1
Hypoproteinemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laparoscopy (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ophthalmoplegia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 | 0 (0) | 0 (0) | 0 (0) | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1
Peritonitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Period 2 High Dose OM (N=95) | Cohort A: Period 2 Low Dose OM (N=95) | Cohort A: Period 3 OM High Dose Continued (N=48) | Cohort A: Period 3 Placebo From High Dose (N=45) | Cohort A: Period 3 OM Low Dose Continued (N=45) | Cohort A: Period 3 Placebo From Low Dose (N=44) | Cohort A: Period 4 Open-label OM (N=178) | Cohort B: Period 2 High Dose OM (N=56) | Cohort B: Period 2 Low Dose OM (N=56) | Cohort B: Period 3 OM High Dose Continued (N=26) | Cohort B: Period 3 Placebo From High Dose (N=28) | Cohort B: Period 3 OM Low Dose Continued (N=27) | Cohort B: Period 3 Placebo From Low Dose (N=26) | Cohort B: Period 4 Open-label OM (N=103) | Cohort C: Period 2 Open-label OM (N=59) | Cohort C: Period 3 OM Dose Continued (N=29) | Cohort C: Period 3 Placebo (N=28) | Cohort C: Period 4 Open-label OM (N=57)
Abdominal pain upper (Gastrointestinal disorders) | 3 | 5 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 4 | 4 | 3 | 0 (0) | 0 (0) | 0 (0) | 16 | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 | 3 | 0 (0) | 0 (0) | 7
Nasopharyngitis (Infections and infestations) | 1 | 4 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 16 | 1 | 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 | 1 | 0 (0) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 7 | 4 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 20 | 0 (0) | 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 | 1 | 1 | 0 (0) | 11
Dizziness (Nervous system disorders) | 9 | 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 | 0 (0) | 0 (0) | 1 | 0 (0)
Headache (Nervous system disorders) | 14 | 7 | 4 | 1 | 3 | 2 | 30 | 5 | 3 | 2 | 0 (0) | 1 | 1 | 18 | 1 | 0 (0) | 0 (0) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 2 | 0 (0) | 1 | 1 | 12 | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 3 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 | 3 | 3 | 0 (0) | 0 (0) | 0 (0) | 11 | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 | 0 (0) | 0 (0) | 0 (0) | 3
Influenza (Infections and infestations) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 | 10 | 0 (0) | 2 | 1 | 0 (0) | 1 | 0 (0) | 4 | 1 | 1 | 1 | 3
Pharyngitis (Infections and infestations) | 4 | 2 | 0 (0) | 3 | 2 | 0 (0) | 7 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 | 0 (0) | 1 | 1 | 24 | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 7 | 3 | 1 | 1 | 5
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 (0) | 0 (0) | 2 | 0 (0) | 4 | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 | 0 (0) | 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 | 0 (0) | 0 (0) | 0 (0) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 | 1 | 0 (0) | 1 | 4
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 0 (0) | 3
Tonsilitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4
Viral infection (Infections and infestations) | 0 (0) | 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3
Pseudohyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5
Proteinurea (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 | 0 (0) | 0 (0) | 0 (0) | 6
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 | 0 (0) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If identified by Daiichi Sankyo Inc.(DSI), any of DSI's confidential information, as defined to the author, shall be deleted. Nothing in our site agreement shall be taken as giving DSI any right of editorial control over any publication prepared by the study site.